CLINICAL TRIAL: NCT00253968
Title: Efficacy and Safety of Eplivanserin 5mg/Day on Sleep Maintenance Insomnia: a 12-week, Multicenter, Randomized, Double-blind, Placebo-controlled Study
Brief Title: Efficacy and Safety of Eplivanserin Treatment for Sleep Maintenance Insomnia
Acronym: GEMS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LTE6217; 2005-003080-23 (EudraCT Number)
Record Dates: First submitted 2005-11-14; First posted 2005-11-15 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Sleep Initiation and Maintenance Disorders; Insomnia
Keywords: Primary Insomnia; Sleeplessness; Early Awakening; Chronic Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — SR 46349B

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eplivanserin (Experimental): Eplivanserin 5 mg/day
  Interventions: Drug: Eplivanserin
- Placebo (Placebo Comparator): Placebo of Eplivanserin 5 mg /day
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Eplivanserin — oral administration
  Other Names: (SR46349)
  Arms: Eplivanserin
Drug: placebo — oral administration
  Arms: Placebo

SUMMARY:
The purpose of the study is to assess efficacy and safety of eplivanserin in the population of patients complaining of sleep maintenance insomnia. The patients suffering from that condition frequently wake up during the night, their sleep is nonrestorative and they suffer from a significant distress or impairment in their daily activities consecutive to insomnia.

DETAILED DESCRIPTION:
12 weeks for each patient (double-blind period) + 1 week of run-in (placebo), and 2 weeks of run-out (placebo)

Total Duration of observation: 15 weeks for each patient

ELIGIBILITY:
Inclusion Criteria:

* Out patients
* Each patient must have primary insomnia in accordance with DSM-IV-TR-Axis I (Diagnostic and Statistical Manual of Mental Disorders- Fourth Edition-Text Revision) criteria
* Based on patient's information, the patient must complain of at least one hour of wakefulness after sleep onset for at least 3 nights per week over the preceding month
* Patient must report impact daytime functioning associated with sleep maintenance insomnia as measured by question 3 of Insomnia Severity Index at screening visit and randomization visit.

Exclusion Criteria:

* Females who are lactating or pregnant
* Woman of childbearing potential with a positive serum beta human chorionic gonadotropin pregnancy test at screening and not using an acceptable form of contraception
* Patients presenting with acute or chronic pain resulting in insomnia
* Patients with history of epilepsy or seizures
* Consumption of xanthine containing beverage (i.e. tea, coffee, or cola) comprising more than 5 glasses/day
* Evidence of any clinically significant, severe, or unstable acute or chronically progressive medical or surgical disorder which may affect patient safety
* BMI >32
* Acute or chronic pain resulting in insomnia
* Patients with current psychiatric disorders according to DSM-IV-TR criteria, mental retardation, or dementia
* Clinically significant and abnormal EKG (QTc interval >=500 msec)
* Positive for hepatitis B or C
* Serious head injury or stroke within 1 year
* Use of OTC (over-the-counter) medications such as valerian root, kava, melatonin, St. John's Wort, or alluna; prescription sleep medications or anxiolytics within 1 week or 5 half-lives
* Participation in another trial within two month before the screening visit
* Use of any substance with psychotropic effects or properties known to affect sleep/wake
* Unable to complete the study questionnaires
* Night shift workers, and individuals who nap 3 or more times per week over the preceding month
* History of:

  * Primary hypersomnia
  * Narcolepsy
  * Breathing-related sleep disorder (such as sleep apnea)
  * Circadian rhythm sleep disorder
  * Parasomnia (somnambulism)
  * Dyssomnia (such as periodic leg movements)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 967 (Actual)
Dates: Start 2005-11; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline of the mean pr-WASO (wake time after sleep onset using patient's sleep questionnaire) | at week 12

SECONDARY OUTCOMES:
Change from baseline of the mean of the FOSQ (Functional Outcome of Sleep Questionnaire) items 1 and 2 (concentration/memory) | at week 12
Change from baseline of the mean of the FOSQ items 4 and 10 (hobby/work) | at week 12

CONTACTS AND LOCATIONS:
Overall Officials: ICD, Study Director — Sanofi
Locations (12):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Buenos Aires, Argentina
- Sanofi-Aventis Administrative Office, Macquarie Park, Australia
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Santiago, Chile
- Sanofi-Aventis Administrative Office, Prague, Czechia
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, México, Mexico
- Sanofi-Aventis Administrative Office, Gouda, Netherlands
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Guildford, United Kingdom